CLINICAL TRIAL: NCT05031754
Title: Assessing SleeP IN Infants With Early-onset Atopic Dermatitis by Longitudinal Evaluation
Brief Title: Assessing SleeP IN Infants With Atopic Dermatitis by Longitudinal Evaluation
Acronym: SPINDLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Collaborators: Wellcome Trust (Other); Health Service Executive, Ireland (Other); Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 223047/Z/21/Z
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis; Sleep Disturbance
MeSH Terms: conditions — Dermatitis, Atopic; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Inflammatory cytokine analysis is being performed by tape stripping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with atopic dermatitis: Infants with atopic dermatitis
- Infants without atopic dermatitis: Infants without atopic dermatitis

SUMMARY:
The SPINDLE study will examine sleep in infants with atopic dermatitis by serial assessment over the first year of life, in comparison to infants without atopic dermatitis. Sleep will be assessed using electroencephalography, actigraphy, and sleep questionnaires.

DETAILED DESCRIPTION:
Infants will be recruited at 6 to 8 months and followed up until 18 months of age. Sleep electroencephalography will be performed at 6 to 8 months. Sleep actigraphy will be performed at 6 to 8 months and 12 months. Infant sleep questionnaires will be completed on a monthly basis, and parental sleep questionnaires will be completed at 6 to 8 months, 9 to 10 months, and 12 months. A neurodevelopmental assessment will be performed at 18 months.

ELIGIBILITY:
Inclusion Criteria:

- Moderate to severe atopic dermatitis

Exclusion Criteria:

* Premature birth (under 37 weeks gestation)
* Severe medical condition (such as epidermolysis bullosa or ichthyosis) at time of enrolment that would complicate assessment for AD or preclude the use of investigational tools, or other major health problems (especially genetic or metabolic) that would have implications for neurodevelopment
* Any medical condition requiring the using of sedating medications (eg antihistamines)

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants under six months of age diagnosed with moderate to severe AD are eligible for the study. Healthy control infants, matched in age, will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Altered macrostructure of sleep from 6 to 12 months measured with parental sleep diaries | 6 months to 12 months
  Measured as decreased sleep efficiency and increased night time awakenings
Altered macrostructure of sleep at 6 and 12 months measured by nocturnal actigraphy | 6 months, 12 months
  Measured as sensor-detected movement

SECONDARY OUTCOMES:
Altered microstructure of sleep at six-eight months using electroencephalography to measure sleep spindle power in rapid eye movement and non-rapid eye movement stages | 6-8 months
  Measured as sleep spindle power and power in rapid eye movement (REM) and non-rapid eye movement (NREM) sleep stages
Parental sleep quality and quality of life measured using the Pittsburgh Sleep Quality Index (PSQI) | 6 months to 12 months
  Measured using standardized questionnaire (PSQI)

OTHER OUTCOMES:
Severity of atopic dermatitis in cases as assessed using SCORAD (SCORing Atopic Dermatitis) | 6 months to 12 months
  Measured using standardized clinical assessment score (SCORAD)
Severity of atopic dermatitis in cases as assessed using the Eczema Area and Severity Index (EASI) | 6 months to 12 months
  Measured using standardized clinical assessment score (EASI)
Severity of atopic dermatitis in cases as assessed using Investigator's Global Assessment scale (IGA) | 6 months to 12 months
  Measured using standardized clinical assessment scores (IGA)
Neurodevelopmental assessment | At 18 months of age (one-off assessment)
  Measured using novel touchscreen app ('Cognitot')

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Boylan, PhD, Principal Investigator — INFANT, University College Cork
Locations (1):
- INFANT, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Connor C, Irvine AD, Murray D, Murphy M, O'B Hourihane J, Boylan G. Study protocol: assessing SleeP IN infants with early-onset atopic Dermatitis by Longitudinal Evaluation (The SPINDLE study). BMC Pediatr. 2022 Jun 18;22(1):352. doi: 10.1186/s12887-022-03382-3. PMID 35717147